CLINICAL TRIAL: NCT06577116
Title: An Open-Label Extension Study Evaluating the Safety, Tolerability, PK, Immunogenicity, and Clinical Response of Multiple Doses of IV AK006 in Subjects With H1 Antihistamine Refractory Chronic Spontaneous Urticaria Completing Study AK006-001
Brief Title: Open-Label Extension Study for Subjects With H1 Antihistamine Refractory Chronic Spontaneous Urticaria Completing Study AK006-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK006-001X
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 720mg of AK006 IV (Experimental): Subjects in this arm will receive 4 doses of 720mg of AK006 via intravenous infusion every 4 weeks.
  Interventions: Drug: AK006 IV

INTERVENTIONS:
Drug: AK006 IV — Formulation for intravenous infusion

SUMMARY:
An open label extension (OLE) study offered to subjects with Chronic Spontaneous Urticaria that have completed the AK006-001 (NCT06072157) Part C referred to as the Main study portion of the study. Qualified subjects will receive up to four doses of the study drug (AK006) through an intravenous infusion every 4 weeks. There is a 16-week follow up period once all the scheduled infusions have been completed. Subjects will be follow for evaluation of safety, tolerability, PK, immunogenicity, and clinical response.

ELIGIBILITY:
Key Inclusion Criteria:

* Enrolled in Part C of Study AK006-001 (NCT06072157) and completed the randomized, double-blind, placebo-controlled treatment period and the Day 99 Visit.
* Acceptable demonstration of tolerance to study drug during the AK006-001 study as determined by the investigator.
* Acceptable demonstration of protocol compliance during the AK006-001 study as determined by the investigator.
* Female subject of childbearing potential and male subject with female partner of childbearing potential must agree to use a highly effective method of contraception with <1% failure rate or abstain from sexual activity from Screening until the end of the study, or for 16 weeks following the last dose of AK006, whichever is longer.

Key Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant while participating in the study.
* Planned use of an approved or investigational therapy to treat CSU other than a single 2nd- or later-generation H1-AH between 1× and 4× the licensed dose and frequency, during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs), treatment-emergent adverse events, serious adverse events, adverse events of special interest, AEs leading to discontinuation | Through study completion, approximately 30 weeks
Incidence of clinically significant abnormal laboratory values, ECGs, and vital signs | Through study completion, approximately 30 weeks

SECONDARY OUTCOMES:
AK006 serum concentrations | Through study completion, approximately 30 weeks
AK006 Anti-drug Antibodies (ADAs) | Through study completion, approximately 30 weeks
  Number of participants with positive or negative AK006-ADAs.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (9):
  - Site 601-004, Birmingham, Alabama
  - Site 601-014, Bakersfield, California
  - Site 601-015, Upland, California
  - Site 601-006, Overland Park, Kansas
  - Site 601-019, Lexington, Kentucky
  - Site 601-011, St Louis, Missouri
  - Site 601-002, Cincinnati, Ohio
  - Site 601-010, El Paso, Texas
  - Site 601-013, Greenfield, Wisconsin
- Canada (5):
  - Site 601-106, Calgary, Alberta
  - Site 601-107, Niagara Falls, Ontario
  - Site 601-108, Toronto, Ontario
  - Site 601-102, Québec, Quebec
  - Site 601-105, Québec, Quebec